CLINICAL TRIAL: NCT02502188
Title: A Phase 1, Multicenter, Randomized, Double-blind, Placebo-controlled, Single and Multiple Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CC-90005 in Healthy Subjects and Subjects With Moderate to Severe Plaque-type Psoriasis
Brief Title: Phase 1 Study of CC-90005 in Healthy Subjects and Subjects With Moderate to Severe Plaque-type Psoriasis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-90005-CP-001
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Parapsoriasis; Healthy Volunteers
Keywords: Healthy Subjects; Severe Plaque Psoriasis; Moderate; Phase 1; Safety; Tolerability; CC-90005
MeSH Terms: conditions — Parapsoriasis; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 - CC-90005 and Placebo (Experimental): CC-90005 or Placebo will be administered orally from low to high dose
  Interventions: Drug: CC-90005; Drug: Placebo
- Part 2 - CC-90005 and Placebo (Experimental): CC-90005 or Placebo will be administered orally from low to high dose
  Interventions: Drug: CC-90005; Drug: Placebo

INTERVENTIONS:
Drug: CC-90005
Drug: Placebo

SUMMARY:
To evaluate the safety, tolerability, and pharmacokinetics of single and multiple doses of CC-90005 in healthy subjects and subjects with moderate to severe plaque-type psoriasis.

DETAILED DESCRIPTION:
This is a 2-part study to be conducted at multiple study centers. Part 1 is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics of CC-90005 following a single oral dose in healthy subjects. During the course of Part 1, each subject will participate in a screening phase, baseline phase(s), treatment phase(s) and a follow up visit. There will be a total of 3 planned cohorts, each of which will consist of a different dose level, with 8 subjects per cohort. In each cohort, 6 subjects will receive a dose of CC 90005 and 2 subjects will receive placebo depending on the randomization schedule. Each cohort will receive a minimum of 2 doses, with one of the cohorts receiving a third dose (up to three study periods per cohort). Administration of study drug at the next higher dose level will not begin until the safety and tolerability of the preceding dose have been evaluated and deemed acceptable by the investigator and sponsor's medical monitor. Part 2 is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics of CC-90005 following multiple oral doses in subjects with moderate to severe plaque-type psoriasis. During the course of Part 2, each subject will participate in a screening phase, a baseline phase, a treatment phase and a follow up visit. There will be a total of 4 planned cohorts, each of which will consist of a different dose level, with 12 subjects per cohort. In each cohort, 9 subjects will receive a dose of CC-90005 and 3 subjects will receive placebo depending on the randomization schedule. It is planned for study drug to be administered twice daily for 28 days. Proposed dose levels in Part 2 may be modified and/or eliminated based on data obtained from Part 1 and/or from previous data obtained in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 (Healthy Subjects)

Subjects must satisfy the following criteria to be enrolled in the study:

1. Female or male subject is ≥ 18 and ≤ 65 years of age at the time of signing the informed consent form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject is in good health as determined by a physical examination at screening.
5. Female subjects of childbearing potential (FCBP) 1 must:

   1. Have two negative pregnancy tests as verified by the Investigator prior to the first dose of Investigational Product (IP). She must agree to ongoing pregnancy testing during the course of the study, and prior to discharge from the clinical site. This applies even if the FCBP subject practices true abstinence from heterosexual contact.
   2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, effective contraception without interruption, during the study (including dose interruptions) and for at least 28 days after discontinuation of IP.

   The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization).
6. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle-stimulating hormone [FSH] level of > 40 IU/L at screening)
7. Male subjects must:

   a. Practice true abstinence (which must be reviewed on a monthly basis and source documented) or agree to use a condom during sexual contact with a pregnant female or FCBP while participating in the study, during dose interruptions and for at least 28 days after discontinuation of IP, even if he has undergone a successful vasectomy.
8. Subject has body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
9. Subject has platelet count, absolute neutrophil count, and absolute lymphocyte count above the lower limit of normal at screening.
10. Subject has liver function tests below the upper limit of normal at screening.
11. For all other clinical laboratory safety test parameters, the subject has results within normal limits or acceptable to the Investigator.
12. Subject is afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 140 mmHg, supine diastolic BP ≥ 50 and ≤ 90 mmHg, and pulse rate ≥ 40 and ≤ 110 bpm at screening.
13. Subject has a normal or clinically-acceptable 12-lead ECG at screening. In addition:

    1. If male, subject has a QTcF value ≤ 430 msec at screening.
    2. If female, subject has a QTcF value ≤ 450 msec at screening.

       * Part 2 (Subjects with Moderate to Severe Plaque-type Psoriasis)

Subjects must satisfy the following criteria to be enrolled in the study:

1. Female or male subject is ≥ 18 and ≤ 70 years of age at the time of signing the ICF.
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject is generally healthy, with the exception of the underlying psoriasis, as determined by medical history review, physical examination, 12-lead ECG, clinical chemistry, hematology, and urinalysis at screening.
5. Subject has a clinical diagnosis of stable moderate to severe plaque-type psoriasis at least 6 months prior to screening, defined as:

   1. PASI score ≥ 12;
   2. BSA ≥ 10%; and
   3. sPGA score ≥ 3.
6. FCBP must:

   1. Have two negative pregnancy tests as verified by the Investigator prior to the first dose of IP. She must agree to ongoing pregnancy testing during the course of the study, and prior to discharge from the clinical site. This applies even if the FCBP subject practices true abstinence from heterosexual contact.
   2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, effective contraception without interruption, during the study (including dose interruptions) and for at least 28 days after discontinuation of IP.

   The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization).
7. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a FSH level of > 40 IU/L at screening)
8. Male subjects must:

   a. Practice true abstinence (which must be reviewed on a monthly basis and source documented) or agree to use a condom during sexual contact with a pregnant female or FCBP while participating in the study, during dose interruptions and for at least 28 days after discontinuation of IP, even if he has undergone a successful vasectomy.
9. Subject is a candidate for photo/systemic therapy. A subject is considered a candidate for photo/systemic therapy if, in the judgment of the Investigator, the subject requires any ultraviolet (UV) radiation or systemic therapy (eg, ultraviolet light B [UVB], psoralens and long-wave ultraviolet radiation [PUVA], methotrexate, cyclosporine, corticosteroids, oral retinoids, mycophenolate mofetil, thioguanine, hydroxyurea, sirolimus, tacrolimus, azathioprine, or approved biological agent) to control psoriasis, whether or not the subject has a history of receiving systemic therapy.
10. Subject has an antitetanus immunoglobulin (Ig) G titer ≥ 0.15 IU/mL to ensure prior exposure of tetanus toxoid (Bingham, 2010).

Exclusion Criteria:

* Part 1 (Healthy Subjects)

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant and relevant medical condition (including but not limited to neurological, gastrointestinal (GI), renal, hepatic, CV, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders), laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject is pregnant or breastfeeding.
5. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or five half-lives of that investigational drug, if known (whichever is longer).
6. Subject has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days prior to the first dose administration.
7. Subject has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days prior to the first dose administration.
8. Subject has used CYP3A inducers and/or inhibitors (including St. John's wort) within 30 days prior to the first dose administration. The Indiana University "Cytochrome P450 Drug Interaction Table" should be utilized to determine inhibitors and/or inducers of CYP3A (http://medicine.iupui.edu/clinpharm/ddis/table.aspx).
9. Subject has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion, eg, bariatric procedure. Appendectomy and cholecystectomy are acceptable.
10. Subject donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
11. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before the first dose administration, or positive drug screening test reflecting consumption of illicit drugs.
12. Subject has a history of alcohol abuse (as defined by the current version of the DSM) within 2 years before the first dose administration, or positive alcohol screen.
13. Subject is known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.
14. Subject smokes > 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
15. Subject had systemic infection within 30 days prior to the first dose administration.
16. Subject has a previous history of autoimmune disease.
17. Subject is part of the clinical staff personnel or a family member of the clinical site staff.

    * Part 2 (Subjects with Moderate to Severe Plaque-type Psoriasis)

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant and relevant medical condition (including but not limited to neurological, GI, renal, hepatic, CV, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major uncontrolled disease), laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject is pregnant or breastfeeding.
5. Subject has known active, current or history of recurrence of bacterial, viral, fungal, mycobacterial, or other infections (including but not limited to tuberculosis [TB] and atypical mycobacterial disease, and herpes zoster), HIV, or any major episode of infection requiring hospitalization or treatment with intravenous or oral antibiotics within 4 weeks prior to screening.
6. Subject completed treatment for mycobacterial infection (ie, TB) at least 3 years prior to screening but lacks documentation.
7. Subject has a positive QuantiFERON-Gold test or two successive indeterminate QuantiFERON-Gold tests at screening. Subjects with a history of TB who have undergone treatment (documented) may be eligible for study entry.
8. Subject has a history of incompletely treated Mycobacterium tuberculosis infection, as indicated by:

   1. Subject's medical records documenting incomplete treatment for Mycobacterium tuberculosis.
   2. Subject's self-reported history of incomplete treatment for Mycobacterium tuberculosis.
9. Subject has any clinically significant findings/abnormalities on chest X-ray at screening.
10. Subject is known to have serum hepatitis or known to be a carrier of HBsAg or HCV Ab, or have a positive result to the test for HIV antibodies at screening.
11. Subject has a history of positive congenital and acquired immunodeficiencies (eg, Common Variable Immunodeficiency [CVID]).
12. Subject has a history of solid tumors and hematologic malignancies. Note: Subjects with a history of squamous or basal cell carcinoma of the skin or cervical intraepithelial neoplasia (CIN) or in situ cervical carcinoma that has been excised and cured > 5 years from screening are eligible for study entry.
13. Subject has psoriasis flare within 4 weeks before screening, defined as a sudden intensification of psoriasis requiring prescribed medical intervention or a diagnosis of erythrodermic, guttate, or pustular psoriasis.
14. Subject has evidence of skin conditions that would interfere with evaluations related to the effect of IP on psoriasis.
15. Subject received topical therapy within 14 days prior to the first dose administration (including but not limited to topical corticosteroids, topical retinoids or vitamin D analog preparations, tacrolimus, pimecrolimus, or anthralin). Exceptions: low potency corticosteroids will be allowed as background therapy for treatment of the face, axillae and groin in accordance with the manufacturers' suggested usage during the course of the study. Subjects with scalp psoriasis will be permitted to use coal tar shampoo and/or salicylic acid scalp preparations on scalp lesions. Eucerin® cream (the standard emollient for this study) will also be permitted for body lesions only. Subjects must not use these treatments within 24 hours prior to each check-in.
16. Subject received systemic therapy for psoriasis within 4 weeks prior to the first dose administration (including but not limited to cyclosporine, corticosteroids, methotrexate, oral retinoids, mycophenolate mofetil, thioguanine, hydroxyurea, sirolimus, tacrolimus, azathioprine, fumaric acid esters, and apremilast).
17. Subject used phototherapy (eg, UVB, PUVA) within 4 weeks prior to the first dose administration.
18. Subject used adalimumab, etanercept, efalizumab or infliximab within 12 weeks prior to the first dose administration.
19. Subject used alefacept omalizumab, rituximab, ustekinumab, briakinumab, or other therapeutic antibody products within 24 weeks prior to the first dose administration.
20. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or five half-lives of that investigational drug, if known (whichever is longer).
21. Subject has a history of alcohol, drug or chemical abuse within 6 months prior to screening.
22. Subject had a major surgery within 8 weeks prior to screening and/or planned major surgery during the entire length of the study.
23. Subject has prolonged sun exposure or uses tanning booths or other UV light sources.
24. Subject received tetanus vaccination within 5 years prior to the first dose administration.
25. Subject self-reports a history of hypersensitivity to any component of TENIVAC® or any other tetanus or diphtheria toxoid-containing vaccine, including hypersensitivity to latex.
26. Subject self-reports any previous unacceptable adverse reaction, ie, extreme hypersensitivity or allergy, to Candida albicans antigen or to a similar product, immunization, or shellfish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-07-17 (Actual); Primary Completion 2015-11-02 (Actual); Study Completion 2015-11-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to 12 months
  Number of participants with adverse events

SECONDARY OUTCOMES:
Pharmacokinetics- Cmax | Up to 28
  Maximum observed plasma concentration
Pharmacokinetics- Tmax | Up to 28
  Time to Cmax (Maximum observed plasma concentration)
Pharmacokinetics- AUC∞ | Up to 28 days
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics- AUCt | Up to 28 days
  Area under the plasma concentration-time curve from time zero to the last quantifiable concentration
Pharmacokinetics- AUC24 | Up to 28 days
  Area under the plasma concentration-time curve from time zero to 24 hours post dose
Pharmacokinetics- AUCτ | Up to 28 days
  Area under the plasma concentration-time curve from time zero to tau (τ), where τ is the dosing interval
Pharmacokinetics- t1/2 | Up to 28 days
  Terminal elimination half-life
Pharmacokinetics- CL/F | Up to 28 days
  Apparent total plasma clearance when dosed orally
Pharmacokinetics- Vz/F | Up to 28 days
  Apparent total volume of distribution when dosed orally, based on the terminal phase
Pharmacokinetics- RAc | Up to 28 days
  Ratio of accumulation
Quality of Life Analysis | Up to Day 36
  Dermatology Life Quality Index will be used to assess quality of life throughout study
Body Surface Area Involvement | Up to Day 36
  Standard body surface area grading scale will be used to assess severity of psoriasis throughout study
Psoriasis Area and Severity Index Scores | Up to Day 36
  Standard psoriasis area and severity index scale will be used to assess severity of psoriasis throughout study
Static Physicians Global Assessment score | Up to Day 36
  Static physicians global assessment score will be used to assess severity of psoriasis throughout study
Effect of CC-90005 on ECG parameters | Up to 50 hours
  12-lead ECGs will be extracted from continuous Holter recordings and used to assess the effect of CC-90005 on ECG parameters

CONTACTS AND LOCATIONS:
Overall Officials: Maria Palmisano, MD, Study Director — Celgene Corporation
Locations (1):
- PPD Development, LP, Austin, Texas, United States